CLINICAL TRIAL: NCT01385475
Title: Efficacy of Resistance Training Guidelines to Improve Function in Older Adults
Brief Title: Resistance Training to Improve Physical Function in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Scott J Strath PhD, University of Wisconsin-Milwaukee
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RTFunction; K01AG025962 (NIH)
Record Dates: First submitted 2011-06-22; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Physical Function
Keywords: Resistance Training; Physical Function; Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control (Experimental)
  Interventions: Behavioral: RT

INTERVENTIONS:
Behavioral: RT — 8 week RT Intervention

SUMMARY:
The primary purpose of this study is to examine the effectiveness of the current resistance training guidelines for older adults proposed by ACSM/AHA to improve physical function in individuals with reduced physical abilities. A randomized controlled intervention trial will be used to compare change in physical function pre- and post-intervention between a treatment group receiving the minimum recommendations of the guidelines and a control group asked not to change their physical activity participation. To better understand the clinical significance of such an occurrence, a secondary purpose was to determine if older adults with reduced physical abilities who adhere to the recommended intervention dosage will experience a change such that they can be reclassified to a more favorable level of functioning. It is hypothesized that the minimum recommended dosage of the guidelines would be sufficient to both improve physical function and improve functional classification in older adults with reduced physical abilities.

ELIGIBILITY:
Inclusion Criteria:

* Older Adults aged >65yrs; reduced physical function

Exclusion Criteria:

* Those with a history of resistance training

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Functionality | 8 weeks
  Change in Short Performance Physical Battery (SPPB) score is used as a measure of functionality. The SPPB consists of three tasks designed to assess gait speed, and ability to rise from a chair and maintain standing balance. This is a common test to assess function, with scores ranging from 0-12. The higher score equates to a better level of function.

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Strath, PhD, Study Director — University of Wisconsin, Milwaukee
Locations (1):
- Physical Activity & Health Research Laboratory, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Gennuso KP, Zalewski K, Cashin SE, Strath SJ. Resistance training congruent with minimal guidelines improves function in older adults: a pilot study. J Phys Act Health. 2013 Aug;10(6):769-76. doi: 10.1123/jpah.10.6.769. Epub 2012 Oct 10. PMID 23074076